CLINICAL TRIAL: NCT06261554
Title: Efficacy and Safety of Low-dose Sesame Oral Immunotherapy in Pediatric Patients: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Low-dose Sesame Oral Immunotherapy in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low-dose sesame OIT
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-02

CONDITIONS: Food Allergy
Keywords: sesame; food allergy; immunotherapy; children
MeSH Terms: conditions — Food Hypersensitivity; SeSAME syndrome | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sesame immunotherapy (Experimental): Children with sesame allergy receiving OIT.
  Interventions: Dietary Supplement: Dietary Supplement: Low dose OIT
- Sesame avoidance (No Intervention): Children with sesame allergy not undergoing OIT.

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Low dose OIT — Following the building-up phase (up to 14 months), patients will receive a daily low dose of sesame paste (300 mg sesame protein) mixed with well-tolerated fruit mousse or bread for 3 months (12 +/- 3 weeks).
  Arms: Sesame immunotherapy

SUMMARY:
It is a randomized, single-center, controlled trial to evaluate the effectiveness of oral immunotherapy with low-dose sesame protein compared with standard treatment (elimination diet) in patients with sesame allergy.

DETAILED DESCRIPTION:
Allergic reactions to sesame can be severe and life-threatening, making it challenging to avoid hidden sources of the allergen.

This pilot study is a randomized controlled trial evaluating the efficacy and safety of oral immunotherapy (OIT) with a low-dose sesame protein in pediatric patients with sesame allergy. The study aims to compare participants undergoing OIT with a maintenance dose of 300mg sesame protein against a control group in a 2:1 randomized allocation. The control group will be recommended a standard treatment, which is a restrictive elimination diet and the use of emergency treatment, including adrenaline, in case of accidental exposure to sesame.

39 participants aged 3-17 with confirmed IgE-mediated sesame allergy will be enrolled into the study. Interventions will be administered once daily for up to 18 months, and the control group will stay under observation for one year.

Primary outcomes include the proportion of participants tolerating a single dose of 4000mg sesame protein during the final oral food challenge. Secondary outcomes assess adverse events, changes in immunological parameters, and the maximum tolerated doses of sesame protein in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 17 years,
* IgE-mediated sesame allergy confirmed with positive skin prick tests with sesame allergens (diameter of the wheal greater than 3mm) and/or specific IgE level greater than 0.35-kilo units of Allergen per liter (kUA/l),
* Allergic reaction to sesame protein during oral food challenge (OFC),
* Signed Informed Consent by parent/legal guardian and patient aged >16 years old,
* Patient's and caregivers' cooperation with the researcher.

Exclusion Criteria:

* No confirmed sesame allergy,
* Negative OFC with sesame protein (maximum dose 4000mg),
* Severe asthma, uncontrolled mild/moderate asthma: forced expiratory volume at one second (FEV1)<80% (under 5. percentile), FEV1/forced vital capacity (FVC)<75% (under 5. percentile), hospitalization due to asthma exacerbation within last 12 months,
* Current oral/sublingual/subcutaneous immunotherapy with other allergens in the first year of immunotherapy,
* Eosinophilic gastroenteritis,
* A history of severe recurrent anaphylaxis episodes,
* Chronic diseases requiring continuous treatment, including heart disease, epilepsy, metabolic diseases, diabetes,
* Medication:

  * oral, daily steroid therapy longer than 1 month within the last 12 months,
  * at least two courses of oral steroid therapy (at least 7 days) within the last 12 months,
  * oral steroid therapy longer than 7 days within the last 3 months,
  * any biological treatment,
  * therapy with β-blockers, angiotensin-converting enzyme (ACE) inhibitors, calcium channel inhibitors,
* Pregnancy,
* No consent to participate in the study,
* Lack of patient or caregiver cooperation.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Tolerance of sesame | Up to 18 months after starting oral immunotherapy
  The proportion of participants who tolerate the single dose of 4000mg sesame protein at the conclusion of the study.

SECONDARY OUTCOMES:
Adverse event | Up to 18 months after starting oral immunotherapy
  Quantity and severity of adverse effect, assessed and compared between groups, divided into 3 categories: mild, moderate and severe reactions
Laboratory data | Up to 18 months after starting oral immunotherapy
  Difference in sesame serum immunoglobulin E (IgE) level and immunoglobulin G4 (IgG4) level, compared between groups at the end of treatment.
Basophil activation test | Up to 18 months after starting oral immunotherapy
  The basophil activation test (BAT) results compared between groups at the end of treatment.
Skin prick test (SPT) | Up to 18 months after starting oral immunotherapy
  Change in skin prick test reactivity to sesame protein from baseline to end of treatment, compared between groups.
Desensitization dose | Up to 18 months after starting oral immunotherapy
  Change in maximum tolerated dose of sesame in oral food challenge before and in the end of treatment, compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices)
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Gupta RS, Warren CM, Smith BM, Blumenstock JA, Jiang J, Davis MM, Nadeau KC. The Public Health Impact of Parent-Reported Childhood Food Allergies in the United States. Pediatrics. 2018 Dec;142(6):e20181235. doi: 10.1542/peds.2018-1235. Epub 2018 Nov 19. Erratum In: Pediatrics. 2019 Mar;143(3):e20183835. doi: 10.1542/peds.2018-3835. PMID 30455345
- [Background] Warren CM, Jiang J, Gupta RS. Epidemiology and Burden of Food Allergy. Curr Allergy Asthma Rep. 2020 Feb 14;20(2):6. doi: 10.1007/s11882-020-0898-7. PMID 32067114
- [Background] Gupta RS, Warren CM, Smith BM, Jiang J, Blumenstock JA, Davis MM, Schleimer RP, Nadeau KC. Prevalence and Severity of Food Allergies Among US Adults. JAMA Netw Open. 2019 Jan 4;2(1):e185630. doi: 10.1001/jamanetworkopen.2018.5630. PMID 30646188
- [Background] Sicherer SH, Warren CM, Dant C, Gupta RS, Nadeau KC. Food Allergy from Infancy Through Adulthood. J Allergy Clin Immunol Pract. 2020 Jun;8(6):1854-1864. doi: 10.1016/j.jaip.2020.02.010. PMID 32499034
- [Background] Dalal I, Goldberg M, Katz Y. Sesame seed food allergy. Curr Allergy Asthma Rep. 2012 Aug;12(4):339-45. doi: 10.1007/s11882-012-0267-2. PMID 22610362
- [Background] Osborne NJ, Koplin JJ, Martin PE, Gurrin LC, Lowe AJ, Matheson MC, Ponsonby AL, Wake M, Tang ML, Dharmage SC, Allen KJ; HealthNuts Investigators. Prevalence of challenge-proven IgE-mediated food allergy using population-based sampling and predetermined challenge criteria in infants. J Allergy Clin Immunol. 2011 Mar;127(3):668-76.e1-2. doi: 10.1016/j.jaci.2011.01.039. PMID 21377036
- [Background] Warren CM, Chadha AS, Sicherer SH, Jiang J, Gupta RS. Prevalence and Severity of Sesame Allergy in the United States. JAMA Netw Open. 2019 Aug 2;2(8):e199144. doi: 10.1001/jamanetworkopen.2019.9144. PMID 31373655
- [Background] Aaronov D, Tasher D, Levine A, Somekh E, Serour F, Dalal I. Natural history of food allergy in infants and children in Israel. Ann Allergy Asthma Immunol. 2008 Dec;101(6):637-40. doi: 10.1016/S1081-1206(10)60228-1. PMID 19119709
- [Background] Nachshon L, Goldberg MR, Levy MB, Appel MY, Epstein-Rigbi N, Lidholm J, Holmqvist M, Katz Y, Elizur A. Efficacy and Safety of Sesame Oral Immunotherapy-A Real-World, Single-Center Study. J Allergy Clin Immunol Pract. 2019 Nov-Dec;7(8):2775-2781.e2. doi: 10.1016/j.jaip.2019.05.031. Epub 2019 May 29. PMID 31150789
- [Background] Begin P, Winterroth LC, Dominguez T, Wilson SP, Bacal L, Mehrotra A, Kausch B, Trela A, Hoyte E, O'Riordan G, Seki S, Blakemore A, Woch M, Hamilton RG, Nadeau KC. Safety and feasibility of oral immunotherapy to multiple allergens for food allergy. Allergy Asthma Clin Immunol. 2014 Jan 15;10(1):1. doi: 10.1186/1710-1492-10-1. PMID 24428859
- [Background] Adatia A, Clarke AE, Yanishevsky Y, Ben-Shoshan M. Sesame allergy: current perspectives. J Asthma Allergy. 2017 Apr 27;10:141-151. doi: 10.2147/JAA.S113612. eCollection 2017. PMID 28490893
- [Background] Brough HA, Caubet JC, Mazon A, Haddad D, Bergmann MM, Wassenberg J, Panetta V, Gourgey R, Radulovic S, Nieto M, Santos AF, Nieto A, Lack G, Eigenmann PA. Defining challenge-proven coexistent nut and sesame seed allergy: A prospective multicenter European study. J Allergy Clin Immunol. 2020 Apr;145(4):1231-1239. doi: 10.1016/j.jaci.2019.09.036. Epub 2019 Dec 20. PMID 31866098
- [Background] Sampson HA, Gerth van Wijk R, Bindslev-Jensen C, Sicherer S, Teuber SS, Burks AW, Dubois AE, Beyer K, Eigenmann PA, Spergel JM, Werfel T, Chinchilli VM. Standardizing double-blind, placebo-controlled oral food challenges: American Academy of Allergy, Asthma & Immunology-European Academy of Allergy and Clinical Immunology PRACTALL consensus report. J Allergy Clin Immunol. 2012 Dec;130(6):1260-74. doi: 10.1016/j.jaci.2012.10.017. No abstract available. PMID 23195525
- [Background] Feuille E, Nowak-Wegrzyn A. Allergen-Specific Immunotherapies for Food Allergy. Allergy Asthma Immunol Res. 2018 May;10(3):189-206. doi: 10.4168/aair.2018.10.3.189. PMID 29676066
- [Derived] Zielinska J, Zagorska W, Krupa-Laska A, Lyzwa K, Lewandowski Z, Kulus M, Grzela K. Efficacy and safety of low-dose sesame oral immunotherapy in paediatric patients: a protocol for a single-centre, randomised controlled trial. BMJ Open. 2024 Aug 12;14(8):e085811. doi: 10.1136/bmjopen-2024-085811. PMID 39134434